CLINICAL TRIAL: NCT05411666
Title: Maintenance Optimization of the Fully Implanted Venous Catheter
Acronym: OTIMACAT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Clinical Academic Center (2CA-Braga) (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: OTIMACAT
Record Dates: First submitted 2022-05-26; First posted 2022-06-09 (Actual); Last update posted 2025-08-15 (Actual); Status verified 2025-08

CONDITIONS: Cancer
Keywords: Central venous catheter
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm 1 (Other): Saline solution maintenance of the Central venous catheter (CVC)
  Interventions: Procedure: Saline solution maintenance of the CVC
- Arm 2 (Experimental): No maintenance of the Central venous catheter (CVC)
  Interventions: Procedure: No maintenance of the CVC

INTERVENTIONS:
Procedure: Saline solution maintenance of the CVC — Saline solution maintenance of the Central venous catheter (CVC) - Celsite IMPLANTOFIX from B|Braun, according to local standard procedures.
  Other Names: Saline solution maintenance
  Arms: Arm 1
Procedure: No maintenance of the CVC — No maintenance of the Central venous catheter (CVC) - Celsite IMPLANTOFIX from B|Braun. Just visual inspection to local site of CVC insertion.
  Other Names: No maintenance
  Arms: Arm 2

SUMMARY:
Central venous catheter (CVC) are intravascular devices used in clinical practice, namely to administer fluid therapy, parenteral nutrition, drugs, blood products, hemodynamic monitoring, also being a gateway to the collection of blood samples or laboratory monitoring.

The fully implanted central venous catheter (CVCTI) is a type of central venous access surgically placed, which is characterized by containing a subcutaneous reservoir that is accessed by puncturing the camera with a blunt needle, widely used in cancer patients. The fully implanted central venous catheter is recommended when there is a need for intermittent vascular access and of long duration.

The maintenance of the CVCTI, as it's the necessity, frequency, and method is subject of some controversy, with discrepancies between the various cancer centers and guidance documents, once they occur several different intervals and maintenance methods.

The objective of this study is to assess the necessity of frequent maintenance of fully implanted central venous catheter, still assuring its viability and holding the same or lower number incidence of complications.

Participants in this study are cancer patients with a CVC fully implanted for chemotherapy, in follow-up phase. Participants will be randomized in one of two arms: Maintenance with saline solution and no maintenance.

ELIGIBILITY:
Inclusion Criteria:

* Patients over 18 years of age.
* Cancer patients, undergoing placement of CVCTI for chemotherapy, in follow-up, who finished chemotherapy up to a maximum period of 10 weeks.
* Eastern Cooperative Oncology Group (ECOG) status of 0 or 1
* Evidence of signed and dated informed consent indicating that the patient has been informed of all relevant aspects of the study and agrees to participate.

Exclusion Criteria:

* Presence of metastases or any other condition that may be an indication for intravenous treatments or additional chemotherapy regimens
* History of CVCTI-related adverse events during the treatment phase
* Patients on anticoagulant medication
* History of thrombophilia
* Pregnancy/Breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 176 (Estimated)
Dates: Start 2020-06-30 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Number of Adverse Events | Time since screening until follow-up visit (on average 20 months)
  The occurrence of any adverse event related to the use of the CVCTI, thus allowing to assess the difference between the 2 groups with as much data as possible.

SECONDARY OUTCOMES:
Occurence of AE related with infectious complications | Time since screening until follow-up visit (on average 20 months)
  The occurrence of adverse events related to infectious complications in the 2 groups.
Occurence of AE related with thrombotic complications | Time since screening until follow-up visit (on average 20 months)
  The occurrence of adverse events related to thrombotic complications of both CVCTI and venous thrombosis in both groups.

CONTACTS AND LOCATIONS:
Overall Officials: Ema Alves, Principal Investigator — Serviço de Hospital de Dia, Hospital de Braga, EPE
Locations (1):
- Serviço de Hospital de Dia, Hospital de Braga, Braga, Portugal